CLINICAL TRIAL: NCT04414735
Title: Impact of Photopheresis in the Prevention of Acute Rejection in Highly Sensitized de Novo Kidney Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Fritz Diekmann, Head of the Experimental Laboratory of Nephrology and Transplantation (LENIT), Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCB/2018/0853
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Kidney Transplant Rejection
Keywords: Kidney Transplant Rejection; photopheresis; Antibody-mediated rejection; Chronic active antibody-mediated rejection
MeSH Terms: interventions — Photopheresis

STUDY DESIGN:
Intervention Model Description: Unicentric, randomized, open study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- Control group (Standard immunosuppression) (No Intervention): 1- Control group (n=15): Standard immunosuppression (Thymoglobulin, Prednisone, Tacrolimus, and Everolimus or Mycophenolate), according to the clinical protocol of the Nephrology and Kidney Transplant Department.
- 2- Treatment group (ECP+Standard immunosuppression) (Experimental): 2- Treatment group (n=15): Extracorporeal photopheresis in combination with standard immunosuppression (Thymoglobulin, Prednisone, Tacrolimus, and Everolimus or Mycophenolate) according to the clinical protocol of the Nephrology and Kidney Transplant Department
  Interventions: Other: Extracorporeal Photopheresis

INTERVENTIONS:
Other: Extracorporeal Photopheresis — Infusion of autologous cellular products exposed to ultraviolet light (UV), in the presence of a photosensitizer. The cellular product is obtained through leucopheresis and its subsequent exposure to 8-methoxypsoralen (8-MOP) and irradiation with UV-A light.
  Arms: 2- Treatment group (ECP+Standard immunosuppression)

SUMMARY:
The aim of the present study is to evaluate the superiority of photopheresis in combination with the standard immunosuppression vs standard immunosuppression alone for the prevention of acute rejection in highly sensitized kidney transplant recipients (cPRA ≥90%).

Unicentric, randomized, open study.

ELIGIBILITY:
Inclusion Criteria:

* Sensitized (cPRA ≥90%) candidates for a deceased-donor kidney transplantation
* Recipients between 18 and 75 years old
* Patients are able to understand and sign informed consent (Annex 1).

Exclusion Criteria:

* Participation in another interventional clinical trial.
* Use of Rituximab or Eculizumab at the time of transplant or in the first 24 hours post-transplant.
* Persons with any dependency on the researcher or employee by the responsible institution or researcher. As well as people detained by legal order.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to first histological rejection in the first year of kidney transplantation. | 1 year after kidney transplantation
  Time to first histological rejection in the first year of kidney transplantation.

SECONDARY OUTCOMES:
Biopsy proved acute rejection | 1 year after kidney transplantation
Glomerular filtrate rate at one year after kidney transplant | 1 year after kidney transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Nephology and Kidney Transplant, Barcelona, Please Select, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaksch P, Knobler R. ECP and solid organ transplantation. Transfus Apher Sci. 2014 Jun;50(3):358-62. doi: 10.1016/j.transci.2014.04.006. Epub 2014 Apr 13. PMID 24768429
- [Background] Heshmati F. Updating ECP action mechanisms. Transfus Apher Sci. 2014 Jun;50(3):330-9. doi: 10.1016/j.transci.2014.04.003. Epub 2014 Apr 13. PMID 24837416
- [Background] Rose EA, Barr ML, Xu H, Pepino P, Murphy MP, McGovern MA, Ratner AJ, Watkins JF, Marboe CC, Berger CL. Photochemotherapy in human heart transplant recipients at high risk for fatal rejection. J Heart Lung Transplant. 1992 Jul-Aug;11(4 Pt 1):746-50. PMID 1498142
- [Background] Barr ML, Meiser BM, Eisen HJ, Roberts RF, Livi U, Dall'Amico R, Dorent R, Rogers JG, Radovancevic B, Taylor DO, Jeevanandam V, Marboe CC. Photopheresis for the prevention of rejection in cardiac transplantation. Photopheresis Transplantation Study Group. N Engl J Med. 1998 Dec 10;339(24):1744-51. doi: 10.1056/NEJM199812103392404. PMID 9845709
- [Background] Barr ML, Baker CJ, Schenkel FA, McLaughlin SN, Stouch BC, Starnes VA, Rose EA. Prophylactic photopheresis and chronic rejection: effects on graft intimal hyperplasia in cardiac transplantation. Clin Transplant. 2000 Apr;14(2):162-6. doi: 10.1034/j.1399-0012.2000.140211.x. PMID 10770423
- [Background] Kirklin JK, Brown RN, Huang ST, Naftel DC, Hubbard SM, Rayburn BK, McGiffin DC, Bourge RB, Benza RL, Tallaj JA, Pinderski LJ, Pamboukian SV, George JF, Marques M. Rejection with hemodynamic compromise: objective evidence for efficacy of photopheresis. J Heart Lung Transplant. 2006 Mar;25(3):283-8. doi: 10.1016/j.healun.2005.10.004. Epub 2006 Jan 25. PMID 16507420
- [Background] Pecoraro Y, Carillo C, Diso D, Mantovani S, Cimino G, De Giacomo T, Troiani P, Shafii M, Gherzi L, Amore D, Rendina EA, Venuta F, Anile M. Efficacy of Extracorporeal Photopheresis in Patients With Bronchiolitis Obliterans Syndrome After Lung Transplantation. Transplant Proc. 2017 May;49(4):695-698. doi: 10.1016/j.transproceed.2017.02.035. PMID 28457374
- [Background] Jaksch P, Scheed A, Keplinger M, Ernst MB, Dani T, Just U, Nahavandi H, Klepetko W, Knobler R. A prospective interventional study on the use of extracorporeal photopheresis in patients with bronchiolitis obliterans syndrome after lung transplantation. J Heart Lung Transplant. 2012 Sep;31(9):950-7. doi: 10.1016/j.healun.2012.05.002. PMID 22884382
- [Background] Kusztal M, Koscielska-Kasprzak K, Gdowska W, Zabinska M, Myszka M, Klak R, Krajewska M, Boratynska M, Szyber P, Chudoba P, Patrzalek D, Klinger M. Extracorporeal photopheresis as an antirejection prophylaxis in kidney transplant recipients: preliminary results. Transplant Proc. 2011 Oct;43(8):2938-40. doi: 10.1016/j.transproceed.2011.08.061. PMID 21996194